CLINICAL TRIAL: NCT05012670
Title: An Open-Label, Single-Dose, Single-Period Study to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-Paxalisib in Healthy Male Subjects
Brief Title: Mass Balance Recovery, Metabolite Profile, and Metabolite Identification of [14C]-Paxalisib in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kazia Therapeutics Limited (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KZA-0084-102; QSC204878 (Other: Quotient Sciences)
Record Dates: First submitted 2021-08-04; First posted 2021-08-19 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Phosphatidylinositol 3-Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-Paxalisib Capsule (Experimental): Subjects will be dosed on the morning of Day 1 following an overnight fast of a minimum of 10 h. Subjects will remain resident in the clinical unit until 168 h post dose (Day 8) and this may be extended up to a maximum of 48 h (i.e., up to Day 10).
  Interventions: Drug: [14C]-Paxalisib Capsule

INTERVENTIONS:
Drug: [14C]-Paxalisib Capsule — Each subject will receive a single dose 15 mg (NMT 3.5 MBq), administered orally in the fasted state with with 240 mL water.
  Other Names: Phosphoinositide 3-kinase (PI3K) Inhibitor

SUMMARY:
Single-centre, open-label, non-randomised study to assess the mass balance recovery, PK, metabolite profile, and metabolite identification of a single oral dose of 14C labelled paxalisib ([14C] Paxalisib) in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males.
2. Aged 30 to 65 years inclusive at the time of signing informed consent.
3. Body mass index (BMI) of 18.0 to 35.0 kg/m2 as measured at screening.
4. Must be willing and able to communicate and participate in the whole study.
5. Must have regular bowel movements (i.e., average stool production of ≥1 and ≤3 stools per day).
6. Must provide written informed consent.
7. Must agree to adhere to the contraception requirements defined in study protocol.

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1.
2. Subjects who are, or are immediate family members of, a study site or sponsor employee.
3. Evidence of current SARS-CoV-2 infection.
4. History of any drug or alcohol abuse in the past 2 years.
5. Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type).
6. A confirmed positive alcohol breath test at screening or admission.
7. Current smokers and those who have smoked within the last 12 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission.
8. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months.
9. Subjects with pregnant or lactating partners.
10. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study.
11. Subjects who have been administered IMP in an ADME study in the last 12 months.
12. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening.
13. Clinically significant abnormal clinical chemistry, haematology, or urinalysis as judged by the investigator (laboratory parameters are listed in study protocol).
14. Confirmed positive drugs of abuse test result (drugs of abuse tests are listed in study protocol)
15. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV) antibody results
16. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <80 mL/min using the Cockcroft-Gault equation.
17. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory disease, neurological, or psychiatric disorder, as judged by the investigator.
18. History of clinically significant GI disease, especially peptic ulceration, GI bleeding, ulcerative colitis, Crohn's Disease, or Irritable Bowel Syndrome.
19. Any history of pre-diabetes, diabetes mellitus (any type), or hyperglycaemia. At screening, fasting blood glucose and HbA1c must be within the normal range.
20. History or presence of significant dermatological disorders or skin rashes, as judged by the investigator.
21. Subject had a QTcF of >450 msec based on ECG at screening or at pre dose, or a history of additional risk factors for Torsades de Pointe (e.g., hypokalaemia, hypomagnesia, a family history of long QT syndrome).
22. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
23. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active.
24. Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood.
25. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day) within 14 days before IMP administration (see Section 11.4). COVID-19 vaccines are accepted concomitant medications, except for within 72 h of dosing. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as determined by the investigator.
26. Subjects who have had a COVID-19 vaccine within 72 h (3 days) before IMP administration.
27. History of GI surgery (with the exception of appendectomy unless it was performed within the previous 12 months).
28. Acute diarrhoea or constipation in the 7 days before the predicted Day 1. If screening occurs >7 days before the Day 1, this criterion will be determined on Day 1. Diarrhoea will be defined as the passage of liquid faeces and/or a stool frequency of greater than 3 times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day.
29. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
To determine the mass balance recovery after a single oral dose of carbon-14 ([14C])-Paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Mass balance recovery of total radioactivity (TR) in all excreta (urine and faeces): CumAe (amount excreted) and Cum%Ae
To provide plasma samples for metabolite profiling and structural identification | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Collection of plasma samples for metabolite profiling, structural identification, and quantification analysis of paxalisib metabolites
To provide urine samples for metabolite profiling and structural identification | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Collection of urine samples for metabolite profiling, structural identification, and quantification analysis of paxalisib metabolites
To provide faecal samples for metabolite profiling and structural identification | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Collection of faecal samples for metabolite profiling, structural identification, and quantification analysis of paxalisib metabolites

SECONDARY OUTCOMES:
To determine the routes and rates of elimination of [14C]-Paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Calculation of Ae, %Ae, CumAe, and Cum%Ae for TR by interval in urine and faeces
To identify the chemical structure of each metabolite accounting for more than 10% (in plasma) of circulating TR or metabolites in excreta (urine and faeces) that account for more than 10% of the administered radioactive dose | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Identification of the chemical structure of each paxalisib metabolite accounting for more than 10% by area under the curve (AUC) of circulating TR in plasma to identify major metabolites, and identification of each metabolite in excreta (urine and faeces) that accounts for more than 10% of the administered radioactive dose
To explore the Cmax pharmacokinetic (PK) parameter of paxalisib following administration of [14C] Paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Assessment of the PK of an oral [14C]-Paxalisib formulation by measurement of paxalisib in plasma including but not limited to Cmax parameter
To explore the Tmax pharmacokinetic (PK) parameter of paxalisib following administration of [14C] Paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Assessment of the PK of an oral [14C]-Paxalisib formulation by measurement of paxalisib in plasma including but not limited to Tmax parameter
To explore the AUC(0-last) and AUC(0-inf) pharmacokinetic (PK) parameter of paxalisib following administration of [14C] Paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Assessment of the PK of an oral [14C]-Paxalisib formulation by measurement of paxalisib in plasma including but not limited to AUC(0-last) and AUC(0-inf) parameter
To explore the Cmax pharmacokinetic (PK) of TR following administration of [14C] Paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Assessment of the PK of an oral [14C]-Paxalisib formulation by measurement of TR in plasma including but not limited to Cmax parameter
To explore the Tmax pharmacokinetic (PK) of TR following administration of [14C] Paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Assessment of the PK of an oral [14C]-Paxalisib formulation by measurement of TR in plasma including but not limited to Tmax parameter
To explore the AUC(0-last) and AUC(0-inf) pharmacokinetic (PK) of TR following administration of [14C] Paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Assessment of the PK of an oral [14C]-Paxalisib formulation by measurement of TR in plasma including but not limited to AUC(0-last) and AUC(0-inf) parameter
To evaluate the extent of distribution of TR into blood cells | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Evaluation of whole blood:plasma concentration ratios for TR
To provide adverse event (AE) safety information for paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  To provide safety information for paxalisib by assessing adverse events.
To provide blood pressure vital sign safety information for paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Measuring and assessing blood pressure in standard clinical units and against reference range.
To provide heart rate vital sign safety information for paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Measuring and assessing heart rate in standard clinical units against reference range.
To provide oral temperature vital sign safety information for paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Measuring and assessing oral temperature in standard clinical units against reference range.
To provide respiratory rate vital sign safety information for paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Measuring and assessing respiratory rate in standard clinical units against reference range .
To provide electrocardiogram (ECG) safety information for paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Determination of standard ECG parameters including but not limited to PR interval, QRS duration, in standard clinical units against reference range
To provide physical examination safety information for paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Assessment of standard clinical whole-body targeted (symptom-driven) physical examination including but not limited to e.g. general appearance, dermatological
To provide hematology laboratory safety testing information for paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Measuring and assessing standard array of hematology parameters (e.g. white blood cell count) in standard clinical unit against reference range.
To provide clinical chemistry laboratory safety testing information for paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Measuring and assessing standard array of clinical chemistry parameters (e.g. cholesterol) in standard clinical unit against reference range

OTHER OUTCOMES:
To assess the urine PK of paxalisib following administration of [14C] Paxalisib | Day 1 to Day 8 (or up to Day 10 if discharge criteria not met at Day 8)
  Determination of [14C] Paxalisib and calculation of Ae (amount excreted), CumAe (cummulative amount excreted), %Ae (fraction of dose excreted) and Cum%Ae (cummulative fraction of dose excreted) as appropriate for paxalisib in urine

CONTACTS AND LOCATIONS:
Overall Officials: Philip Evans, MBChB, MRCS, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No